CLINICAL TRIAL: NCT05854810
Title: Single Versus Double Frozen Embryo Transfer in PCOS Patients
Brief Title: Frozen Embryo Transfer in PCOS Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Walid Mohamed Elnagar, Assistant professor of gynecology, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZU-IRB 10066/27-11-2022
Record Dates: First submitted 2023-05-02; First posted 2023-05-11 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PCOS Patient (Active Comparator)
  Interventions: Procedure: fertilized embryo Insertion
- Male factor infertility (Active Comparator)
  Interventions: Procedure: fertilized embryo Insertion

INTERVENTIONS:
Procedure: fertilized embryo Insertion — insertion of single fertilized embryo through IVF
  Arms: PCOS Patient
Procedure: fertilized embryo Insertion — insertion of double fertilized embryo through IVF
  Arms: Male factor infertility

SUMMARY:
Polycystic ovarian syndrome (PCOS) is condition characterized by being complex, familial and polygenetic metabolic condition with heterogeneous involvement of several genes in the hypothalamic-pituitary-gonadal axis. PCOS is the most incident endocrine-metabolic syndrome that is characterized by hyperandrogenemia, menstrual irregularities, and/or small cysts in one or both ovaries and could be considered as the main cause of female infertility.

Assisted reproductive technologies (ART) were defined by the American Center for Disease Control as any fertility-related treatments where eggs or embryos are manipulated. In vitro fertilization involves the transfer of fresh embryos, however, the freeze-all strategy that entails cryopreservation of all embryos to be transferred subsequently in un-stimulated cycle to guard against the negative effects of controlled ovarian stimulation on the endometrium and to minimize the risk of ovarian hyper-stimulation syndrome. Intracytroplasmatic sperm injection (ICSI) is a common procedure used to improve reproductive results, even among couples without male factor infertility.

However, there are several points of controversy in the fields of ART traditionally, multiple embryo transfer strategy was used to increase the chance for getting a baby, however, multiple pregnancy is a common complication for this strategy with subsequent adverse fetal, maternal and neonatal outcomes. Also, the developmental stage of embryos at time of transfer; cleavage versus blastocyst was a matter of debit, but giving the chance for in-vitro maturation to the stage of blastocyst increased the possibility of getting good quality embryo to be transferred. However, the exaggeration of prolongation of the in-vitro duration appeared as a trend, but recent studies found no advantages for transfer of D7 or D6 blastocyst over D5 blastocyst transfer (BT).

ELIGIBILITY:
Inclusion Criteria:

* Infertile women fulfilling at least two of the Rotterdam criteria for diagnosis of PCOS;
* aged 20-35 years;
* had body mass index (BMI) of less than 35 kg/m2;
* mild hirsutism on Ferriman-Gallwey (FG) visual scoring system;
* their hormonal profile of serum AMH >4.5, FSH <5.85 LH>5.39;
* had no previous attempts of ICSI were included in the study.

Exclusion Criteria:

* Patients who were out of the predetermined age range and BMI;
* had uterine abnormalities;
* hydrosaplnix;
* recurrent miscarriage;
* medical diseases interfering with or being complicated by occurrence of pregnancy;
* cases requiring ICSI with TESE samples;
* had obesity-inducing endocrinopathy
* severe symptomatizing hypovitaminosis or maintained on hormonal contraception within the last 6 months before inclusion in the study, were excluded from the study.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 271 (Actual)
Dates: Start 2019-06-07 (Actual); Primary Completion 2022-03-05 (Actual); Study Completion 2022-07-25 (Actual)

PRIMARY OUTCOMES:
the live birth rate (LBR) after SBT and DBT | 9 months

CONTACTS AND LOCATIONS:
Locations (1):
- Zagazig University, Zagazig, Ash Sharqia Governorate, Egypt